CLINICAL TRIAL: NCT06299137
Title: Ultrasound Guided Serratus Anterior Plane Block in ED Patients With Rib Fractures,
Brief Title: Ultrasound Guided Serratus Anterior Plane Block in ED Patients With Rib Fractures
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Leland Perice, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RE2022-0000000349; RE2022-0000000349 (Other Grant/Funding Number: Society of Academic Emergency Medicine)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Rib Fractures; Pain Acute; Regional Anesthesia; Opioid Use
Keywords: rib fractures; regional anesthesia; Opioid use; acute pain
MeSH Terms: conditions — Rib Fractures; Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistants who collect the data will be blinded to which arm of the study the participants are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Usual care. No changes made or recommended to patients randomized to the control arm.
- Intervention arm (Undergoes SAPB) (Experimental): Patients randomized to this arm will receive the Serratus Anterior Plane block.
  Interventions: Procedure: Serratus Anterior Plane Block; Drug: Ropivacaine injection

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — Patients who undergo randomization to the intervention arm will undergo the Serratus Anterior Plane Block.
  Arms: Intervention arm (Undergoes SAPB)
Drug: Ropivacaine injection — For the Serratus Anterior Plane Block, Ropivacaine will be used as the anesthetic.
  Other Names: Ropivacaine
  Arms: Intervention arm (Undergoes SAPB)

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the Serratus Anterior Plane Block in patients with rib fractures. The main questions it aims to answer are:

* Determine if UG-SAPB results in an improved pain, incentive spirometry, and cough ability (PIC) score when compared to usual care over the first five hours.
* Evaluate if UG-SAPB results in fewer opioid medications administered when compared to usual care over the first 24 hours.

Participants will undergo the Serratus Anterior Plane. Researchers will compare this to usual care to see if this intervention improves pulmonary function and reduces opioid requirements for ED patients with rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Radiology confirmed anterior or lateral rib fractures either on X-ray or chest computed tomography CT
* pain score of 5/10.
* Patients must be able to verbalize how much pain they are having on an 11-point Numeric Rating Pain Scale
* perform an incentive spirometry and be able to cough on command

Exclusion Criteria:

* isolated rib fractures that do not include ribs T3-T9
* penetrating trauma, pregnancy
* requiring immediate surgical or procedural intervention
* known allergy to amide-type local anesthetics
* have a painful distracting injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
PIC Score | 5 hours
  Determine if the SAPB results in an improved pain, incentive spirometry, and cough ability (PIC) score when compared to usual care over the first five hours. The PIC score is a scoring system that can be measured serially in patients with rib fractures to assess pulmonary function and to prognosticate clinical outcomes.

SECONDARY OUTCOMES:
Total oral morphine equivalents over the first 24 hours | 24 hours
  Evaluate if UG-SAPB results in fewer opioid medications administered when compared to usual care over the first 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this point as to where and how IPD will be shared for this pilot study.

REFERENCES:
- [Background] Paul S, Bhoi SK, Sinha TP, Kumar G. Ultrasound-Guided Serratus Anterior Plane Block for Rib Fracture-Associated Pain Management in Emergency Department. J Emerg Trauma Shock. 2020 Jul-Sep;13(3):208-212. doi: 10.4103/JETS.JETS_155_19. Epub 2020 Sep 18. PMID 33304071
- [Background] Kring RM, Mackenzie DC, Wilson CN, Rappold JF, Strout TD, Croft PE. Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Improves Pain Control in Patients With Rib Fractures. J Ultrasound Med. 2022 Nov;41(11):2695-2701. doi: 10.1002/jum.15953. Epub 2022 Feb 2. PMID 35106815
- [Background] Lin J, Hoffman T, Badashova K, Motov S, Haines L. Serratus Anterior Plane Block in the Emergency Department: A Case Series. Clin Pract Cases Emerg Med. 2020 Jan 21;4(1):21-25. doi: 10.5811/cpcem.2019.11.44946. eCollection 2020 Feb. PMID 32064417
- [Background] Thiruvenkatarajan V, Cruz Eng H, Adhikary SD. An update on regional analgesia for rib fractures. Curr Opin Anaesthesiol. 2018 Oct;31(5):601-607. doi: 10.1097/ACO.0000000000000637. PMID 30020155
- [Background] Sarode AL, Ho VP, Pieracci FM, Moorman ML, Towe CW. The financial burden of rib fractures: National estimates 2007 to 2016. Injury. 2021 Aug;52(8):2180-2187. doi: 10.1016/j.injury.2021.05.027. Epub 2021 May 19. PMID 34059325